CLINICAL TRIAL: NCT00638716
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose, Phase II Study to Evaluate the Efficacy and Safety of 3 Months of Weekly Injections of CJC-1134-PC in Patients With Type 2 Diabetes Mellitus on Metformin Monotherapy
Brief Title: A Study to Evaluate the Efficacy and Safety of CJC-1134-PC in Patients With Type 2 Diabetes Mellitus Who Are Currently on Metformin Monotherapy
Acronym: DM200-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ConjuChem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM200-101
Record Dates: First submitted 2008-03-13; First posted 2008-03-19 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, incretins, GLP-1, HbA1c, metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 12 weekly doses of 1.5 mg CJC-1134-PC
  Interventions: Drug: CJC-1134-PC
- 2 (Experimental): 4 weekly doses of 1.5 mg CJC-1134-PC followed by 8 weekly doses of 2.0 mg CJC-1134-PC
  Interventions: Drug: CJC-1134-PC
- 3 (Placebo Comparator): 12 weekly doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CJC-1134-PC — 1.5 or 2.0 mg CJC-1134-PC
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
This is a multicenter, randomized, placebo-controlled, double-blind, Phase II study.

The objective of this study is to evaluate the efficacy and safety of 12 weeks of treatment with CJC-1134-PC in patients with type 2 diabetes mellitus who are currently on metformin monotherapy.

ELIGIBILITY:
Major Inclusion Criteria:

* BMI: 27 to 45 kg/m2
* Stable Type 2 diabetes mellitus for at least 3 months, as defined by the Investigator
* Stable life-style, i.e. diet & physical activity, as determined by the Investigator
* Stable metformin daily dose ≥1000 mg for at least 3 months
* Glycosylated hemoglobin (HbA1c) at screening ≥ 7.1% and ≤ 11%

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ConjuChem Biotechnologies Inc., Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.5 mg CJC-1134-PC: 12 weekly doses of 1.5 mg CJC-1134-PC
  CJC-1134-PC: 1.5 mg CJC-1134-PC
- 1.5 or 2.0 mg CJC-1134-PC: 4 weekly doses of 1.5 mg CJC-1134-PC followed by 8 weekly doses of 2.0 mg CJC-1134-PC
  CJC-1134-PC: 1.5 or 2.0 mg CJC-1134-PC
- Placebo: 12 weekly doses of placebo
  Placebo: Placebo
Period: Overall Study
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo
Started | 50 | 52 | 58
Completed | 43 | 37 | 46
Not Completed | 7 | 15 | 12

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 57 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.46) | 55.1 (12.24) | 57.2 (13.05) | 55.9 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 28 | 30 | 79
  Male | 28 | 21 | 27 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 5 | 17
  Not Hispanic or Latino | 45 | 41 | 52 | 138
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 4 | 5 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 7 | 25
  White | 34 | 33 | 36 | 103
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Reduction of HbA1c From Baseline
Description: Change from Baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Percent (%)
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 44 | 38 | 47
Percent (%) | -0.85 (0.883) | -0.80 (0.827) | -0.46 (0.744)

2. Secondary Outcome: Reduction in FPG From Baseline
Description: Change from Baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 42 | 38 | 45
mg/dL | -13.48 (34.579) | -18.76 (36.736) | -10.06 (34.137)

3. Secondary Outcome: Reduction in Fasting Body Weight From Baseline
Description: Change from Baseline
Time Frame: Screening and Day 85
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo
Number analyzed (Participants) | 44 | 38 | 46
kg | -1.98 (2.438) | -1.25 (2.106) | -1.58 (2.374)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | 1.5 mg CJC-1134-PC | 1.5 or 2.0 mg CJC-1134-PC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/57
Other Adverse Events (participants affected / at risk) | 36/49 | 30/49 | 34/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1.5 mg CJC-1134-PC (N=49) | 1.5 or 2.0 mg CJC-1134-PC (N=49) | Placebo (N=57)
Nausea (Gastrointestinal disorders) | 11 | 15 | 9 — Most common AEs
Diarrhea (Gastrointestinal disorders) | 6 | 6 | 3 — Most common AEs
Vomiting (Gastrointestinal disorders) | 6 | 2 | 2 — Most common AEs
Injection site bruising (General disorders) | 0 | 0 | 3 — Most common AEs
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 — Most common AEs
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 — Most common AEs
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3 — Most common AEs
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 0 — Most common AEs
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 — Most common AEs
Headache (Nervous system disorders) | 5 | 2 | 9 — Most common AEs
Dizziness (Nervous system disorders) | 2 | 2 | 4 — Most common AEs
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 — Most common AEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes